CLINICAL TRIAL: NCT02133625
Title: A Phase I Study of Pioglitazone and Carboplatin in Patients With Advanced Solid Tumors
Brief Title: A Study of Pioglitazone and Carboplatin in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, James Cleary, MD, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-096
Record Dates: First submitted 2014-02-09; First posted 2014-05-08 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Advanced Solid Tumor; Metastatic Solid Tumor
Keywords: Advanced solid tumor; Metastatic solid tumor
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Carboplatin; Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pioglitazone and Carboplatin (Experimental): MTD Determination
  * Pioglitazone: 45 mg Once Daily by mouth,Cycle 1Days 1-28; Subsequent cycles: Days 1-21
  * Carboplatin:6 AUC IV 60 minute infusion (or per institutional policy) Cycle 1: Day 8; Subsequent cycles: Day 1
  Interventions: Drug: carboplatin; Drug: pioglitazone
- MTD Expansion Carboplatin and Pioglitazone (Experimental): MTD Expansion:
  * Carboplatin alone on cycle 1, day 1.
  * Pioglitazone Over days 15-21 of the cycle pioglitazone will be administered alone.
  * On cycle 2, day 1, both carboplatin and pioglitazone will be administered. Cycle 2 and onward are 21-day cycles, with pioglitazone administered once daily and carboplatin administered once every 3 weeks
  Interventions: Drug: carboplatin; Drug: pioglitazone

INTERVENTIONS:
Drug: carboplatin
  Other Names: Paraplatin; CBDCA
Drug: pioglitazone
  Other Names: Actos

SUMMARY:
The proposed investigation is a Phase 1 trial to determine the safety, tolerability, and maximum tolerated dose (MTD) of the combination of pioglitazone ( and carboplatin patients with advanced or metastatic solid malignancies.

DETAILED DESCRIPTION:
* In Part I of the study, the maximum tolerated dose (MTD) will be determined. During part I, Cycle 1, days 1-28, pioglitazone will be administered once daily. On cycle 1, day 8, the first dose of carboplatin will be administered. On cycle 2, day 1, both carboplatin and pioglitazone will be administered. Cycles 2 and onward are 21-day cycles, with pioglitazone administered once daily and carboplatin administered once every 3 weeks. Part I of the study will end when the MTD has been determined in a minimum of 6 patients.
* In Part II of the trial, an MTD Expansion Cohort may be utilized to further characterize the safety profile and pharmacodynamics of the drug. Patients in the MTD Expansion Cohort will receive carboplatin alone on cycle 1, day 1. Over days 15-21 of the cycle pioglitazone will be administered alone. On cycle 2, day 1, both carboplatin and pioglitazone will be administered.

Cycle 2 and onward are 21-day cycles, with pioglitazone administered once daily and carboplatin administered once every 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignancy that is not curable with standard approaches and where carboplatin is appropriate therapy.
* During Part I of the trial (MTD determining phase), measurable or evaluable disease is acceptable. For Part II of the trial (expanded cohort) only, participants must have measurable disease by RECIST criteria version 1.1.
* Participants enrolled in Part II of the trial (expanded cohort) must have disease that is amenable to biopsy with reasonable safety and also be willing to undergo at least two serial tumor biopsies for correlative biomarker investigation as defined in Section 8.2.2.
* Any number of prior therapies are permitted. Prior carboplatin is allowed. Patients who have documented allergy to carboplatin may receive carboplatin with desensitization.

  * Age ≥18 years old.
  * ECOG performance status ≤ 1 (Appendix A).
  * Participants must have normal organ and marrow function as defined below:

    * Absolute neutrophil count ≥1,500/L
    * Hematocrit ≥ 27
    * Platelets ≥100,000/L
    * Total bilirubin within normal institutional limits
    * AST (SGOT)/ALT (SGPT)≤ 2.5 X institutional upper limit of normal
    * Creatinine within normal institutional limits or creatinine clearance ≥ 60 mL/min/1.73 m2 for subjects with creatinine levels above institutional normal.
* Able to swallow oral medication.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

Participants who exhibit any of the following conditions at screening will not be eligible for admission into the study.

* Subjects who have been treated with standard chemotherapy or molecularly targeted agents within the past 3 weeks prior to trial first drug administration.
* Subjects who were receiving experimental therapies must wait 3 weeks from their last dose prior to enrolling. Subjects treated with nitrosoureas or mitomycin C cannot be enrolled until 6 weeks has elapsed since their last treatment.
* Extensive prior radiotherapy on more than 25% of the bone marrow, or prior bone marrow/stem cell transplantation. Prior radiation for local disease management is allowed if last fraction was completed at least 4 weeks prior to trial entry.
* Subjects who have undergone a major surgical procedure within the 6 weeks prior to trial entry.
* History of untreated central nervous system (CNS) metastases. Subjects with a history of prior treated brain metastasis are eligible provided that 1 month following treatment they are stable by CT scan without evidence of cerebral edema, and have no requirements for corticosteroids.
* Diabetic patients who are currently requiring oral hypoglycemic agents or insulin therapy.
* Patients who are currently receiving rosiglitazone or pioglitazone, or who have received dosing with any other agent known to be a PPAR agonist within 3 months prior to study entry.
* Left ventricular ejection fraction ≤ 50% on ECHO or MUGA
* Uncontrolled concomitant illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or nursing women.
* Known HIV positivity, active hepatitis C, or active hepatitis B.
* Patients with ≥ CTCAE Grade 2 peripheral neuropathy.
* Subjects with a known history of gastrointestinal disorder (such as partial esophageal, gastric, small or large bowel obstruction), surgery or malabsorption that could potentially impact the swallowing or the absorption of the study drug.
* Patients taking CYP2C8 inhibitors and inducers (rifampin, gemfibrozil, trimethoprim, montelukast, and quercetin) are excluded from the trial.
* Other significant disease that in the Investigator's opinion would exclude the subject from the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2011-08; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
MTD of pioglitazone and carboplatin | Baseline, 6 Weeks
  To determine the safety, tolerability, and MTD of the combination of pioglitazone (dosed orally once daily at conventional FDA-approved doses) and carboplatin (dosed IV every 3 weeks) in patients with advanced or metastatic solid malignancies. The trial will describe the toxicities of this regimen based on CTCAE. In addition, using RECIST criteria, will look at preliminary anti-tumor activity

SECONDARY OUTCOMES:
Plasma Concentration-time Profiles | 5 minutes pre dosing, at 15 min and 30 min after beginning the infusion, 2 min before the end of the approximately 60 min infusion, and at approximately 30 min, 1 h, 2 h, 4 h, 6 h, and 24 h after the end of the infusion
  The Wilcoxon Signed Rank test will be used to determine whether the addition of pioglitazone (at cycle 2) affects carboplatin pharmacokinetics and pharmacodynamics (assessed during cycle 1 of the MTD cohort). The Wilcoxon Signed Rank test will be used to determine whether the addition of pioglitazone (at cycle 2) affects carboplatin pharmacokinetics and pharmacodynamics (assessed during cycle 1 of the MTD cohort).
Induction Rate of metallothionein expression and DNA damage by carboplatin in the absence or presence of pioglitazone. | Day 2
  To assess induction of metallothionein expression and DNA damage by carboplatin in the absence or presence of pioglitazone. In depth, molecular analysis measuring protein levels of tumor biopsy specimen will be performed to look for molecular predictors of response
Anti-Tumor Response and Progression Rate | Baseline, ≥ 4 Weeks
  To assess preliminary anti-tumor activity of the combination of pioglitazone and carboplatin. We will use RECIST criteria to measure the response rate.

CONTACTS AND LOCATIONS:
Overall Officials: James Cleary, MD, PhD, Principal Investigator — Dana Farber Cancer Instiute
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts